CLINICAL TRIAL: NCT04250883
Title: Low Pressure Pneumoperitoneum and Deep Neuromuscular Blockade Versus Standard Laparoscopy During RARP to Improve the Quality of Recovery and Immune Homeostasis; Study Protocol for a Randomized Controlled Study
Brief Title: Low Pressure Pneumoperitoneum and Deep Neuromuscular Block vs. Standard During RARP to Improve Quality of Recovery; a Randomized Controlled Study.
Acronym: RECOVER-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: NL72780.091.20; 2020-000411-79 (EudraCT Number)
Record Dates: First submitted 2020-01-29; First posted 2020-01-31 (Actual); Results first posted 2025-02-05 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2022-04

CONDITIONS: Quality of Life; Postoperative Complications; Acute Pain; Immune System Tolerance
MeSH Terms: conditions — Postoperative Complications; Acute Pain

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group: Low Impact laparoscopy (Experimental): low impact laparoscopy (low pressure (8 mmHg) and deep NMB (PTC 1-2)
  Interventions: Other: Low intra-abdominal pressure; Other: Deep neuromuscular blockade (NMB)
- Control group: Standard laparoscopy (Active Comparator): standard laparoscopy (standard pressure (14 mmHg) and moderate NMB (TOF 1-2)
  Interventions: Other: Standard intra-abdominal pressure; Other: Moderate neuromuscular blockade (NMB)

INTERVENTIONS:
Other: Low intra-abdominal pressure — 8 mmHg
  Arms: Experimental group: Low Impact laparoscopy
Other: Deep neuromuscular blockade (NMB) — Deep NMB (PTC1-2)
  Arms: Experimental group: Low Impact laparoscopy
Other: Standard intra-abdominal pressure — 14 mmHg
  Arms: Control group: Standard laparoscopy
Other: Moderate neuromuscular blockade (NMB) — Moderate NMB (TOF 1-2)
  Arms: Control group: Standard laparoscopy

SUMMARY:
Intra-abdominal pressure (IAP) needed to create sufficient workspace during laparoscopic surgery affects the surrounding organs with ischemia-reperfusion injury and a systemic immune response. This effect is related to postoperative recovery, pain scores, opioid consumption, bowel function recovery, morbidity and possibly mortality. In clinical practice standard pressures of 12-16mmHg are applied instead of the lowest possible IAP, but accumulating evidence shows lower pressure pneumoperitoneum (PNP) (6-8mmHg) to be non-compromising for sufficient workspace, when combined with deep neuromuscular blockade (NMB) in a vast majority of patients. Therefore, low impact laparoscopy, meaning low pressure PNP facilitated by deep NMB, could be a valuable addition to Enhanced Recovery After Surgery (ERAS) Protocols.

The use of low pressure PNP may also reduce hypoxic injury and the release of DAMPs and thereby contributing to a better preservation of innate immune function which may help to reduce the risk of infectious complications.

The participants will be randomly assigned to one of the experimental groups with low impact laparoscopy or one of the control groups with standard laparoscopy.

DETAILED DESCRIPTION:
Intra-abdominal pressure (IAP) needed to create sufficient workspace during laparoscopic surgery affects the surrounding organs with ischemia-reperfusion injury and a systemic immune response. This effect is related to postoperative recovery, pain scores, opioid consumption, bowel function recovery, morbidity and possibly mortality. Therefore, low impact laparoscopy, meaning low pressure PNP facilitated by deep NMB, could be a valuable addition to Enhanced Recovery After Surgery (ERAS) Protocols.

The use of low pressure PNP may also reduce hypoxic injury and the release of DAMPs and thereby contributing to a better preservation of innate immune function which may help to reduce the risk of infectious complications.

The participants will be randomly assigned to the experimental group 1: low impact laparoscopy (low pressure (8 mmHg) and deep NMB (PTC 1-2)); 8 mmHg IAP after trocar introduction for perfusion measurement or the experimental group 2: low impact laparoscopy (low pressure (8 mmHg) and deep NMB (PTC 1-2)); 12 mmHg IAP after trocar introduction for perfusion measurement, or control group 1: standard laparoscopy (standard pressure (12 mmHg) and moderate NMB (TOF 1-2)); 8 mmHg IAP after trocar introduction for perfusion measurement, or control group 2: standard laparoscopy (standard pressure (12 mmHg) and moderate NMB (TOF 1-2)); 12 mmHg IAP after trocar introduction for perfusion measurement.

ICG injection will take place with starting pressure to quantify parietal peritoneum perfusion, and a parietal peritoneal biopsy will be taken. At the end of surgery, a second parietal peritoneum biopsy will be taken.

NB: After introduction of the camera trocar, insufflation of carbon dioxide is titrated to an IAP of 8mmHg in group A and C, and 14 mmHg in group B and D. After placement of the last trocar the injection of ICG and video registration of peritoneum will take place, and a peritoneal biopsy will be taken. There after surgery will take place with an IAP of 14mmHg in the control groups (C and D), and an IAP of 8mmHg in the experimental groups (A and B). In the control groups (C and D)

Pre- and postoperative a few questionnaires will be taken and blood withdrawals to evaluate the quality of recovery, and the immune response.

ELIGIBILITY:
Inclusion Criteria:

* - Age ≥ 18 years
* Undergoing elective robot assisted radical prostatectomy (RARP)
* Obtained informed consent

Exclusion Criteria:

* Laparoscopic radical prostatectomy without robot assistance
* Insufficient control of the Dutch language to read the patient information and to fill out de questionnaires
* Neo-adjuvant chemotherapy
* Chronic use of analgesics or psychotropic drugs
* Use of NSAID's shorter than 5 days before surgery
* Severe liver- or renal disease
* Neuromuscular disease
* Hyperthyroidism or thyroid adenomas
* Deficiency of vitamin K dependent clotting factors or coagulopathy
* Planned diagnostics or treatment with radioactive iodine < 1 week after surgery
* Indication for rapid sequence induction
* BMI >35kg/m2
* Known of suspected hypersensitivity to ICG, sodium iodide, iodine, rocuronium or sugammadex
* Use of medication interfering with ICG absorption as listed in the summary of product characteristics (SPC); anticonvulsants, bisulphite compounds, haloperidol, heroin, meperidine, metamizol, methadone, morphium, nitrofurantoin, opium alkaloids, phenobarbital, phenylbutazone, cyclopropane, probencid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2020-12-24 (Actual); Primary Completion 2021-12-09 (Actual); Study Completion 2022-03-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michiel Warle, Dr., Principal Investigator — Radboud University Medical Center
Locations (1):
- Canisius Wilhelmina ziekenhuis, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No
All data will be analyzed for publication. After that it belongs to Radboud umc where other researchers of Radboud umc may or may not include this database to their study. But there will be no active sharing

REFERENCES:
- [Result] Reijnders-Boerboom GTJA, Jacobs LMC, Helder LS, Panhuizen IF, Brouwer MPJ, Albers KI, Loonen T, Scheffer GJ, Keijzer C, van Basten JA, Warle MC. Recovery and immune function after low pressure pneumoperitoneum during robot-assisted radical prostatectomy: a randomised controlled trial. BJU Int. 2024 Sep;134(3):416-425. doi: 10.1111/bju.16397. Epub 2024 May 24. PMID 38784993
- See also: Publication of results in BJU international — https://pubmed.ncbi.nlm.nih.gov/38784993/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This blinded, randomized controlled trial was performed at the Canisius Wilhelmina Hospital in Nijmegen. Patients with at least stage T1c prostate cancer scheduled for RARP were randomized to the experimental group with low IAP (8 mmHg) facilitated by deep NMB (PTC 1-2) or the control group with standard IAP (14 mmHg) with moderate NMB (TOF 1-2).
  From December 2020 to December 2021, 236 patients were assessed for eligibility and 97 were included for randomization.
Pre-assignment Details: 139 patients were excluded of which; 29 did not meet inclusion criteria, 99 declined to participate and 11 did not response on invitation.
Groups:
- Experimental Group: Low Impact Laparoscopy: the use of low intra-abdominal pressure (8 mmHg), and deep neuromuscular blockade (PTC1-2)
- Control Group: Standard Laparoscopy: The use of standard intra-abdominal pressure (14 mmHg) and moderate neuromuscular blockade (TOF 1-2)
Period: Overall Study
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Started | 47 | 50
Quality of Recovery Questionnaire at 3 Months | 46 | 50
Completed | 46 (Primary endpoint- quality of recovery: n=46 (lost to follow-up n=1) Secondary endpoints: 1) Ex vivo cytokine responsiveness n=47, 2) parietal perfusion measures n=39 (unclear time of injection n=4, technical problems n=4)) | 50 (Primary endpoint- quality of recovery: n=50 Secondary endpoints: 1) Ex vivo cytokine responsiveness n=50, 2) parietal perfusion measures n=40 (unclear time of injection n=6, technical problems n=4))
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental Group: Low Impact Laparoscopy: Using low intra-abdominal pressure (8 mmHg) and deep neuromuscular blockade (PTC1-2)
- Control Group: Standard Laparoscopy: Using standard intra-abdominal pressure (14 mmHg) and moderate neuromuscular blockade (TOF 1-2)
- Total: Total of all reporting groups
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy | Total
Number analyzed (Participants) | 46 | 50 | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.9 (6.6) | 67.9 (5.1) | 66.4 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 46 | 50 | 96
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 46 | 50 | 96
Body Mass Index (kg/m2) [Mean (Standard Deviation); unit: kg/m2] | 26.6 (2.9) | 27.4 (3.2) | 27.0 (3.0)
American Society of Anesthesiologist classification [Count of Participants; unit: Participants] — ASA 1: Normal healthy patient ASA 2: Patient with mild systemic disease ASA 3: Patient with severe systemic disease
  Participants
    ASA 1 | 22 | 15 | 37
    ASA 2 | 23 | 31 | 54
    ASA 3 | 1 | 4 | 5
Comorbidity [Count of Participants; unit: Participants]
  Cardiovascular: Yes | 22 | 32 | 54
  Cardiovascular: No | 24 | 18 | 42
  Pulmonal: Yes | 2 | 9 | 11
  Pulmonal: No | 44 | 41 | 85
  Neurologic: Yes | 1 | 2 | 3
  Neurologic: No | 45 | 48 | 93
  Diabetic: Yes | 5 | 3 | 8
  Diabetic: No | 41 | 47 | 88
  Renal impairment: Yes | 0 | 0 | 0
  Renal impairment: No | 46 | 50 | 96
  Liver impairment: Yes | 0 | 1 | 1
  Liver impairment: No | 46 | 49 | 95
Tumor characteristics - Risk stratification [Count of Participants; unit: Participants] — Low risk: Tumor is confined to the prostate, PSA is <10 and grade group 1 (Gleason 6). including "slow-growing" tumors with < 3 biopsy tissue samples with cancer cells.
  Intermediate risk: Tumor is confined to the prostate, PSA is between 10 and 20, or grade group 2 or 3 (Gleason 7).
  High risk: Tumor extends outside the prostate, PSA >20, or grade group 4 or 5 (Gleason 8 to 10). Including very aggressive tumors where the tumor has extended into the seminal vesicles (T3b) the rectum or bladder (T4), or multiple biopsy samples with high grade cancer cells.
  Participants
    Low | 9 | 9 | 18
    Intermediate | 28 | 30 | 58
    High | 9 | 11 | 20
Tumor characteristics - Prostate cancer classification [Count of Participants; unit: Participants] — T1 The tumour can't be felt during a DRE or seen with an imaging test. The tumour is found by needle biopsy in one or both sides of the prostate.
  T2 The tumour can be felt by your doctor during a DRE and can be seen on an imaging test. Cancer is only in the prostate.
  T3 The tumour has broken through the outside layer of the prostate gland.
  Participants
    T1c | 21 | 23 | 44
    T2a-c | 19 | 20 | 39
    T3a-c | 5 | 4 | 9
    Unknown | 1 | 3 | 4
Tumor characteristics -Gleason score [Count of Participants; unit: Participants] — Pathologist based; Gleason score ranging in case of cancer from 6-10. A lower score is the lowest grade cancer.
  6: only individual discrete well-formed glands 7: predominantly well-formed glands with lesser component poorly-formed/fused/cribiform glands 8: predominantly poorly-formed/fused/cribiform glands with a lesser component of well-formed glands 9-10: lacks gland formation with or without poorly-formed/fused/cribiform gland.
  Participants
    Score 6 | 10 | 11 | 21
    Score 7 | 30 | 32 | 62
    Score 8 | 3 | 4 | 7
    Score 9 | 3 | 3 | 6
Tumor characteristics - ISUP score [Count of Participants; unit: Participants] — ISUP score based on pattern of Gleason score as determined by pathologist ISUP 1: gleason score <6 and 6 ISUP 2: Gleason score 3+4 =7 ISUP 3: Gleason score 4+3 =7 ISUP 4: Gleason score 4+4 =8 ISUP 5: Gleason score 9 and 10
  Participants
    1 | 10 | 11 | 21
    2 | 23 | 25 | 48
    3 | 8 | 7 | 15
    4 | 3 | 4 | 7
    5 | 3 | 3 | 6
Tumor characteristic - Prostate Cancer specific antigen levels (ng/ml) [Mean (Standard Deviation); unit: ng/ml] | 55.13 (40.4) | 61.74 (47.1) | 58.5 (43.9)
Operation - Pelvic lymph node dissection [Count of Participants; unit: Participants]
  Yes | 21 | 21 | 42
  No | 25 | 29 | 54

OUTCOME MEASURES:

1. Primary Outcome: Quality of Recovery - 40 Items Questionnaire Score (QoR-40)
Description: 40 points (minimum: extremely poor quality of recovery) to 200 points (maximum: excellent quality of recovery)
Time Frame: at postoperative day 1
Measure: Mean (Standard Deviation); unit: score on a scale of 200
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Number analyzed (Participants) | 46 | 50
score on a scale of 200 | 162.7 (21.5) | 167.6 (23.0)
Statistical Analysis 1: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; Test type: Superiority; p = 0.54, Chi-squared, Corrected; for age

2. Primary Outcome: Quality of Recovery - 40 Items Questionnaire Score (QoR-40)
Description: 40 points (minimum: extremely poor quality of recovery) to 200 points (maximum: excellent quality of recovery)
Time Frame: day 12 after surgery
Measure: Mean (Standard Deviation); unit: score on a scale of 200
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Number analyzed (Participants) | 46 | 50
score on a scale of 200 | 179.1 (15.8) | 180.0 (15.1)
Statistical Analysis 1: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; Test type: Superiority; p = 0.97, Chi-squared, Corrected; for age

3. Primary Outcome: Quality of Recovery - 40 Items Questionnaire Score (QoR-40)
Description: 40 points (minimum: extremely poor quality of recovery) to 200 points (maximum: excellent quality of recovery)
Time Frame: Pre-operative
Measure: Mean (Standard Deviation); unit: score on a scale of 200
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Number analyzed (Participants) | 46 | 50
score on a scale of 200 | 186.6 (8.7) | 186.8 (11.5)

4. Secondary Outcome: Health Status With Short Form Survey (SF-36)
Description: Total score on a scale of 0-100 points. The lower the score the more disability. The higher the score the less disability.
Time Frame: Measure pre-operative, on day 12 and at 3 months after surgery
Measure: Mean (Standard Deviation); unit: score on a scale (0-100)
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Number analyzed (Participants) | 46 | 50
score on a scale (0-100)
  Pre-operative | 81.1 (12.1) | 81.8 (11.5)
  12 days postoperative | 61.5 (14.1) | 64.3 (18.7)
  3 months postoperative | 73.7 (15.9) | 77.9 (15.5)
Statistical Analysis 1: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; Test type: Superiority; p = 0.64, Chi-squared, Corrected — At 12 days postoperative; for age
Statistical Analysis 2: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; Test type: Superiority; p = 0.38, Chi-squared, Corrected — At 3 months postoperative; for age

5. Secondary Outcome: Chronic Pain With McGill Pain Questionnaire (MPQ)
Description: Pain Rating index with a range from 0 (no pain) to 78 (severe pain)
Time Frame: 3 months after surgery
Population: 43 participants in de experimental group, and 45 participants in the control group fulfilled the questionnaire. Only 6 participants per group had pain at 3 months after surgery.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Number analyzed (Participants) | 6 | 6
score on a scale | 7.3 (5.0) | 5.7 (9.9)
Statistical Analysis 1: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; Count of patients with or without pain at 3 months postoperative; Test type: Superiority; p = 0.84, Chi-squared, Corrected; For age
Statistical Analysis 2: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; Number of Words Chosen; Test type: Superiority; p = 0.89, ANCOVA; Correction for age
Statistical Analysis 3: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; Pain Rating index; Test type: Superiority; p = 0.98, ANCOVA; Correction for age

6. Secondary Outcome: Operating Conditions
Description: surgical conditions with L-SRS 0 (extremely poor work field) to 5 (excellent work field)
Time Frame: During operation for up to 8 hours
Measure: Mean (Standard Deviation); unit: score on a scale of 0-5
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Number analyzed (Participants) | 46 | 50
score on a scale of 0-5 | 4.9 (0.3) | 4.9 (0.3)
Statistical Analysis 1: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; Test type: Superiority; p = 0.9, ANCOVA; Correction for age

7. Secondary Outcome: Pain Score With NRS
Description: pain scores with NRS 0 (no pain) to 10 (severe pain)
Time Frame: Preset timepoints during hospital stay (1hr, 6hrs, 12hrs, day1), up to 3 days maximum. No measurements after discharge to home.
Population: Patients where in most cases discharged from the hospital on postoperative day 1
Measure: Mean (Standard Deviation); unit: score on a scale of 10
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Number analyzed (Participants) | 46 | 50
score on a scale of 10
  1hour postoperative | 4.1 (2.3) | 3.9 (2.2)
  6hours postoperative | 2.3 (1.1) | 2.3 (1.4)
  12hours postoperative | 2.3 (1.3) | 2.2 (1.4)
  Postoperative day 1 | 1.9 (1.5) | 2.0 (1.4)
Statistical Analysis 1: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; At 1 hour; Test type: Superiority; p = 0.68, ANCOVA; Correction for age
Statistical Analysis 2: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; At 6 hours; Test type: Superiority; p = 0.91, ANCOVA; Correction for age
Statistical Analysis 3: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; Test type: Superiority; p = 0.73, ANCOVA; Correction for age
Statistical Analysis 4: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; Test type: Superiority; p = 0.77, ANCOVA; Correction for age

8. Secondary Outcome: Postoperative Nausea and Vomiting (PONV)
Description: Presence of symptoms yes/no
Time Frame: During hospital stay up to 3 days
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Number analyzed (Participants) | 46 | 50
Participants
  1hour postoperative: Yes | 1 | 0
  1hour postoperative: No | 45 | 50
  Postoperative day 1: Yes | 8 | 4
  Postoperative day 1: No | 38 | 46
Statistical Analysis 1: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; At 1 hour; Test type: Superiority; p = 0.63, ANCOVA; Correction for age
Statistical Analysis 2: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; At postoperative day 1; Test type: Superiority; p = 0.19, ANCOVA; Correction for age

9. Secondary Outcome: Analgesia Use
Description: Cumulative opioid use in morphine equivalent (in mg)
Time Frame: During hospital stay up to 3 days
Measure: Mean (Standard Deviation); unit: mg 'Morphine equivalent'
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Number analyzed (Participants) | 46 | 50
mg 'Morphine equivalent'
  1hour postoperative | 6.2 (5.9) | 5.9 (4.8)
  Postoperative day 1 | 1.3 (3.4) | 0.9 (2.1)
Statistical Analysis 1: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; At 1 hour; Test type: Superiority; p = 0.89, ANCOVA; Correction for age
Statistical Analysis 2: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; At postoperative day 1; Test type: Superiority; p = 0.49, ANCOVA; Correction for age

10. Secondary Outcome: Hospital Stay
Description: length of hospital stay in days
Time Frame: from admission up to 3 days
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Number analyzed (Participants) | 46 | 50
Days | 1.3 (0.7) | 1.24 (0.48)
Statistical Analysis 1: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; Test type: Superiority; p = 0.42, ANCOVA; Correction for age

11. Secondary Outcome: Complications
Description: Postoperative complications scored by Clavien Dindo classification; grade 0 (no deviation from ideal) grade 5 (death of patient)
Time Frame: Day of surgery untill 30days after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Number analyzed (Participants) | 46 | 50
Participants
  Total: Yes | 8 | 10
  Total: No | 38 | 40
  Grade 1: Yes | 4 | 1
  Grade 1: No | 42 | 49
  Grade 2: Yes | 4 | 6
  Grade 2: No | 42 | 44
  Grade 3: Yes | 0 | 2
  Grade 3: No | 46 | 48
  Grade 4: Yes | 0 | 1
  Grade 4: No | 46 | 49
  Grade 5: Yes | 0 | 0
  Grade 5: No | 46 | 50
Statistical Analysis 1: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; Of Total complications within 30 days postoperative; Test type: Superiority; p = 0.92, ANCOVA; Correction for age

12. Secondary Outcome: Perfusion Index of the Parietal Peritoneum
Description: time to maximal intensity in seconds. (extracted from video registration).
Time Frame: From ICG injection, up to 20 seconds
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Number analyzed (Participants) | 39 | 40
seconds
  time to maximal intensity | 48.9 (8.5) | 53.2 (10.2)
  Delta minimal and maximal intensity | 194.4 (41.2) | 169.7 (62.8)
Statistical Analysis 1: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; Time to maximal intensity; Test type: Superiority; p = 0.098, ANCOVA; correction for age
Statistical Analysis 2: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; Angle from minimal to maximal intensity; Test type: Superiority; p = 0.008, ANCOVA; correction for age
Statistical Analysis 3: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; Delta between minimal and maximal intensity; Test type: Superiority; p = 0.042, ANCOVA; correction for age

13. Secondary Outcome: Immune Response Represented by IL-10
Description: IL-10 response upon whole blood LPS stimulation
Time Frame: Pre-operative, postoperative day 1 and 12
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Number analyzed (Participants) | 47 | 50
pg/ml
  preoperative | 6.43 (15.76) | 7.25 (12.45)
  postoperative day 1 | 11.72 (15.45) | 13.94 (17.01)
  postoperative day 12 | 7.24 (15.55) | 8.89 (13.98)
Statistical Analysis 1: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; postoperative day 1; Test type: Superiority; p = 0.35, ANCOVA; Correction for age
Statistical Analysis 2: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; at postoperative day 12; Test type: Superiority; p = 0.52, ANCOVA; Correction for age

14. Secondary Outcome: Immune Response Represented by IL-6
Description: IL-6 response upon whole blood LPS stimulation
Time Frame: Pre-operative, postoperative day 1 and 12
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Number analyzed (Participants) | 47 | 50
pg/ml
  preoperative | 6.60 (22.83) | 8.67 (19.45)
  postoperative day 1 | 20.07 (27.37) | 24.38 (26.67)
  postoperative day 12 | 8.26 (22.9) | 11.95 (20.98)
Statistical Analysis 1: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; at postoperative day 1; Test type: Superiority; p = 0.99, ANCOVA; correction for age
Statistical Analysis 2: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; At postoperative day 12; Test type: Superiority; p = 0.30, ANCOVA; Correction for age

15. Other Pre Specified Outcome: Duration of Surgery
Description: in minutes
Time Frame: 0-350minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Number analyzed (Participants) | 46 | 50
minutes | 198.6 (51.5) | 183.9 (58.7)
Statistical Analysis 1: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; Test type: Superiority; p = 0.42, ANCOVA; Correction for age

16. Other Pre Specified Outcome: Duration of Pneumoperitoneum
Description: in minutes
Time Frame: 0-350 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Number analyzed (Participants) | 46 | 50
minutes | 176.9 (48.3) | 159.8 (56.4)
Statistical Analysis 1: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; Test type: Superiority; p = 0.3, ANCOVA; Correction for age

17. Other Pre Specified Outcome: Estimated Blood Loss
Description: during operation time in ml
Time Frame: During operation
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Number analyzed (Participants) | 46 | 50
ml | 312.8 (333.6) | 214.4 (229.1)
Statistical Analysis 1: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; Test type: Superiority; p = 0.33, ANCOVA; Correction for age

18. Post Hoc Outcome: Complications Based on Infection
Description: patient count
Time Frame: 0-50 patients
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Number analyzed (Participants) | 8 | 10
Participants
  Yes | 5 | 10
  No | 3 | 0
Statistical Analysis 1: Comparison: Experimental Group: Low Impact Laparoscopy vs Control Group: Standard Laparoscopy; Test type: Superiority; p = 0.018, ANCOVA; Correction for age

19. Secondary Outcome: Chronic Pain With McGill Pain Questionnaire (MPQ)
Description: Number of words Chosen according the user manual of the questionnaire
Time Frame: 3 months after surgery
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: number of words describing the pain
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Number analyzed (Participants) | 6 | 6
number of words describing the pain | 3.2 (3.9) | 4.2 (2.5)

20. Secondary Outcome: Perfusion Index of the Parietal Peritoneum
Description: Angle minimal to maximal, calculated from the slope of ICG fluorescence intensity (extracted from video registration).
Time Frame: From ICG injection, up to 20 seconds
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
Number analyzed (Participants) | 39 | 40
Degrees | 82.2 (2.6) | 78.5 (7.9)

ADVERSE EVENTS:
Time Frame: From operation up to 3 months postoperative
Description: according definitions of clinicaltrials.gov
Arm/Group | Experimental Group: Low Impact Laparoscopy | Control Group: Standard Laparoscopy
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/47 | 2/50
Other Adverse Events (participants affected / at risk) | 0/47 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Experimental Group: Low Impact Laparoscopy (N=47) | Control Group: Standard Laparoscopy (N=50)
Small abces in smal pelvic with paralytic ileus (Infections and infestations) | 0 (0) | 1 (1)
Blow out kidney (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
For limitations and caveats we would like to refer you to the publication in BJU International: https://bjui-journals.onlinelibrary.wiley.com/doi/full/10.1111/bju.16397

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/83/NCT04250883/Prot_SAP_000.pdf
  • Informed Consent Form (2020-07-02): https://cdn.clinicaltrials.gov/large-docs/83/NCT04250883/ICF_001.pdf